CLINICAL TRIAL: NCT01087515
Title: Development and Validation of Magnetic Cell Separations Techniques Using a Good Manufacturing Practice (GMP) Grade Manufacturing Process for Clinical Applications and Generation of Pre-clinical Data
Brief Title: Pilot Study for Cell Based Therapies in Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Prof. Dr. Norbert Krug, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09/11 PILOCELL
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood donation (Other)
  Interventions: Other: Blood donation

INTERVENTIONS:
Other: Blood donation — In experimental part 1 to generate preclinical data 250 ml of blood will be donated at day 1 by 10 subjects to induce allergen presenting cells (APCs).
  In experimental part 2 to transfer the isolation of pDC or TREGs to a GMP (good manufacturing Practice) compliant clinical grade isolation system, leukapheresis will be performed with the blood from 5 subjects.
  In experimental part 3 for potency testing of the clinical grade isolation system of pDC or TREGs, 250 ml of blood will be collected at day 1 from 3 subjects.

SUMMARY:
The aim of this study is to investigate the immunomodulatory potential of Isolated Plasmacytoide Dendritic Cells (pDCs) and Regulatory T-cells (TREGs) isolated with clinical grade magnetic bead isolations techniques (MACS®) on the antigen presenting cell-induced proliferation of lymphocytes after allergen uptake in an in vitro cell culture system.

DETAILED DESCRIPTION:
pDCs as well as TREGs will be co-incubated with generated allergen presenting cells, lymphocytes, and allergen. For in vitro experimentation immune cells will be collected from blood of grass mix or house dust mite sensitized atopic/asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects suffering from allergic rhinitis and/or allergic asthma against timothy grass pollen (phleum pratense) and/or house dust mite.
* age 18-60 years,
* Nonsmokers or smokers with a history of less than 1 pack years who have not smoked within the last 12 months.
* Positive skin prick test for timothy grass pollen (phleum pratense) and/or house dust mile within 12 months
* Able and willing to give written informed consent
* Hemoglobin ≥135 g/l
* Hematocrit ≥ 0,40
* Body weight ≥ 50 kg and Body Mass Index (BMI) within the range 19-32 kg/m²

Exclusion Criteria:

* History of lower respiratory tract infection and /or exacerbation of asthma within four weeks prior to the informed consent visit
* Febrile illness within four week before the trial examination
* Administration of oral, injectable, or dermal corticosteroids within the last 8 weeks or intranasal and/or inhaled corticosteroids within the last 4 weeks.
* Intake of methylxanthines, antihistamines, antileukotrienes, oral cromolyn sodium, or oral nedocromil sodium
* Past or present disease, which as judged by the investigator, may affect the outcome of this trial. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease, or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Specific immunotherapy (SIT) within the last two years prior to screening
* Participation in another clinical trial 30 days prior to enrollment
* Donation of more than 500 ml of blood in the preceding 9 weeks before the trial-examination
* Hemoglobin below the normal lower limit
* History of drug and/or alcohol abuse or dependence within 12 months of the trial
* Risk of non-compliance with trial procedures
* Suspected inability to understand the protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial
* Patient is tested human immunodeficiency virus (HIV)-1/2Ab, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV-Ab) positive

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Purity of MACS® and CliniMacs® BDCA-4 positive isolated plasmcytoid dendritic cells: Percentage of CD123/BDCA-2 expressing cells

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Krug, MD, Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine